CLINICAL TRIAL: NCT01916330
Title: Development of Pharmacokinetics Model in Pregnancy Women and Fetus
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SNUHOB-PK1
Record Dates: First submitted 2013-07-29; First posted 2013-08-05 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Preterm Labor; Preterm Premature Rupture of Membrane (PPROM)
MeSH Terms: conditions — Obstetric Labor, Premature; Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Pharmacokinetics analysis and development of pharmacokinetics model in pregnancy women and fetus

ELIGIBILITY:
Inclusion Criteria:

* 20 <= age < 50
* pregnant women who were administered intramuscular dexamethasone (ex) preterm labor)
* pregnant women who were administered PO clarithromycin (ex) PPROM/intrauterine infection or inflammation)

Exclusion Criteria:

* who deny the study entrance
* who administered study drug before transfer to tertiary hospital

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: preterm labor, PPROM in pregnant women from tertiary university hospital
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2014-02-24 (Actual)

PRIMARY OUTCOMES:
Analysis of drug concentration | Day 1 after delivery
  drug (dexamethasone, clarithromycin)

CONTACTS AND LOCATIONS:
Overall Officials: Joong Shin Park, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea